CLINICAL TRIAL: NCT03163862
Title: Granulocyte Stimulating Factor (G-CSF) to Increase the Rate of Implantation Success in IVF Patients in Preferable Preceptive Endometrium Scroe
Brief Title: G-CSF Administration in IVF in a Preferable Preceptive Endometrium Score
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istishari Arab Hospital (Other)
Collaborators: Salem Abu Khyzaran (Unknown); Nizam Najeeb (Unknown)
Responsible Party: Principal Investigator, Areej Khatib, Pathology & clinical labs head department, Istishari Arab Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0001
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-06

CONDITIONS: Women Infertility
Keywords: IVF
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Patients treated with infusion of PLACEBO (saline solution) from the day of embryo transfer through the day of beta hCG test
  Interventions: Drug: Saline Solution
- G-CSF group (Experimental): Patients treated with G-CSF if the biopsy adhesive score 1-3 only, by Endometrial scratching and adhesive factor scoring on day 21-24 cycle prior to IVF//or day 3 of IVF cycle not planned before.
  The dose of G-CSF is 300 µg by trans cervical intrauterine route administered at the oocyte retrieval day, Ans subcutaneous 300µg G-CSF on the day of embryo transfer
  Interventions: Procedure: Endometrial scratch; Drug: G-CSF administration
- Comparative group (Sham Comparator): patients not treated with G-CSF after scratching if the biopsy adhesive score 4 only
  Interventions: Procedure: Endometrial scratch

INTERVENTIONS:
Procedure: Endometrial scratch — the intervention group, endometrial biopsy will be performed with a pipelle de Cornier® (Laboratoires Prodimed, Neully-En-Thelle, France). The pipelle was introduced gently through the cervix up to the uterine fundus. the examiner applied regular back-and-forth movements (2-4 cm) during a period of 30 s. The obtained specimens will be sent for histology evaluation.
  Arms: Comparative group; G-CSF group
Drug: G-CSF administration — 1- 300 µg trans cervical intrauterine of G-CSF was administered at the oocyte retrieval day, subcutaneous 300 micrograms G-CSF on the day of embryo transfer
  Arms: G-CSF group
Drug: Saline Solution — saline infusion every day from the day of embryo transfer through the day of beta HCG test
  Arms: Placebo

SUMMARY:
This is a controlled preminary trial intended to increase the implantation rate of IVF cycles, by using more than one known procedure, endometrial scratching, evaluating the status of the adhesive factors as αVβ3 integrin, L-selectin ligand MECA-79, E-cadherin and ICAM-1, as a determinant for intervention by G-CSF, according to a score that can be done on a small sample obtained during scratching, then give G-CSF for the scores less than 4 intrauterine and subcutaneously.

DETAILED DESCRIPTION:
Placebo: CONTROL patients treated with PLACEBO (saline solution) from the day of embryo transfer through the day of beta hCG test Drug& scratching CONTROL saline infusion every day from the day of embryo transfer through the day of beta HCG test Other Name: SALINE INFUSION Experimental: G-CSF group patients treated with G-CSF if the biopsy adhesive score 1-3 only

1. Endometrial scratching and adhesive factor score, day 21-24 cycle prior to IVF//0rv day 3 of IVF cycle not planned before.
2. Drug &scratching : G-CSF group

1- 300 µg trans cervical intrauterine of G-CSF was administered at the oocyte retrieval day, 2- subcutaneous 300 micrograms G-CSF on the day of embryo transfer Comparative group patients not treated with G-CSF after scratching if the biopsy adhesive score 4 only

Scratching only :

Patients undergoing scratching on day 21-24 of prior IVF cycle/ and on day 5 of IVF cycle with biopsy score of 4.

ELIGIBILITY:
Inclusion Criteria:

* ALL Women aged < 40 years who would be submitted to oocyte retrieval and embryo transfer IN IVF cycle.

Exclusion Criteria:

* • contraindications for G-CSF treatment (sickle cell disease, chronic neutropenia, known past or present malignancy, renal insufficiency, upper respiratory infection, pneumonia, and congenital fructose intolerance)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women aged < 40 years who would be submitted to oocyte retrieval and embryo transfer
Enrollment: 100 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-06-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy per women randomized | 4 weeks
  pregnancy diagnosed by ultrasonographic visualisation of one or more gestational sacs, including ectopic pregnancy

SECONDARY OUTCOMES:
setting a score of precepative endometrium | 12 months
  Evaluation of the endometrial biopsy and setting a receptive score/ adhesive factors of the endometrium

IPD SHARING:
Plan to Share IPD: Undecided